CLINICAL TRIAL: NCT01609452
Title: MONICA-SC: A Randomized, Double-Blind, Placebo-Controlled Phase 2/3 Study to Evaluate the Efficacy, Safety and Tolerability of Blisibimod (A-623) Administration in Subjects With Immune Thrombocytopenic Purpura (ITP)
Brief Title: MONICA-SC: A Study to Evaluate the Efficacy, Safety and Tolerability of Blisibimod (A-623) Administration in Subjects With ITP
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-ITP3321
Record Dates: First submitted 2012-05-23; First posted 2012-06-01 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Immune Thrombocytopenic Purpura; Idiopathic Thrombocytopenic Purpura
Keywords: Immune Thrombocytopenic Purpura; Idiopathic Thrombocytopenic Purpura; Chronic ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — AMG623 peptibody

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Blisibimod (Experimental)
  Interventions: Biological: Blisibimod
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Blisibimod
  Other Names: A-623
  Arms: Blisibimod
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and tolerability of blisibimod when administered on top of standard-of-care to subjects with Immune Thrombocytopenic Purpura (ITP).

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years of age(male or female).
2. Diagnosis of ITP according to the guidelines of the American Society of Hematology (ASH) and British Committee for Standards in Hematology.
3. Platelet counts at Screening of 30 billion/L or less for subjects not on ITP medication, or 50 billion/L or less for subjects receiving stable background ITP medication.

Exclusion Criteria:

1. Subjects who have had a splenectomy for any reason.
2. Currently receiving high-dose ITP medications, eltrombopag, romiplostim, rituximab, or investigational therapeutic agents.
3. Nursing or pregnant.
4. Active infection requiring hospitalization or treatment with parenteral antibiotics within the past 60 days.
5. Any known history of bone marrow stem cell disorder.
6. Active hepatitis B, active hepatitis C or a documented history of HIV, hepatitis B, or hepatitis C.
7. Liver disease.
8. Malignancy within the past 5 years.
9. History of active tuberculosis (TB) or history of TB infection.
10. Subject has not yet completed at least 3 months or 5 half-lives (whichever is longer) since ending other investigational study.
11. History of congenital immunodeficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Achievement of a durable platelet response of 50 billion platelets per liter or higher over the last weeks of treatment. | 24 weeks

SECONDARY OUTCOMES:
Achievement of a durable platelet count of 50 billion platelets per liter or higher over the last weeks of treatment under conditions of decreased concomitant steroid medication. | 24 weeks
Achievement of a transient improvement in platelet count of 50 billion platelets per liter or higher at any 4 weeks of the treatment period. | 24 weeks
Change in background corticosteroid dose. | baseline to 24 weeks
Percentage of subjects requiring rescue therapy. | 24 weeks
Time to treatment failure. | 24 weeks
Change in bleeding risk. | baseline to 24 weeks
Safety profile (AEs, vitals signs, labs) | 24 weeks
Biomarker changes from baseline. | baseline to 24 weeks